CLINICAL TRIAL: NCT07271043
Title: Evaluating the Efficacy of High-Protein Diabetes Specific Formula (HP-DSF) on Body Composition in Overweight/Obese Patients With Type 2 Diabetes Treated With Incretin Mimetic Drugs
Brief Title: Nutrition+: Effect of a High-Protein Diabetes Formula on Body Composition in Type 2 Diabetes Patients Treated With Incretin Mimetics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000322
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants will be instructed to drink two HP-DSF shakes (Protality Base or Ensure Max Protein by (Experimental)
  Interventions: Dietary Supplement: protein supplement
- Participants in this control group will follow the regular standard of diabetes care (No Intervention)

INTERVENTIONS:
Dietary Supplement: protein supplement — HP-DSF shakes (Protality Base or Ensure Max Protein by Abbott Nutrition)
  Arms: Participants will be instructed to drink two HP-DSF shakes (Protality Base or Ensure Max Protein by

SUMMARY:
A randomized clinical study to assess the efficacy of a high-protein diabetes specific formula (HPDSF) on lean muscle mass in overweight and obese patients with type 2 diabetes who are initiating treatment with incretin-mimetic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18-75 years of age
2. Subject was diagnosed with type 2 diabetes at least 3 months prior to screening
3. Subject is about to start treatment with an IMD, a GLP-1 receptor agonist (RA) alone or a dual GLP-1/GIP RA. These treatments include either semaglutide (Ozempic®, Wegovy®), tirzepatide (Mounjaro®, Zepbound®), or dulaglutide (Trulicity®)
4. Body mass index (BMI) is ≥ 25 kg/m2

Exclusion Criteria:

1. Subject has type 1 diabetes mellitus
2. Subject with estimated glomerular filtration rate <60 milliliters/minute/1.73 m²,
3. Urine albumin-to-creatinine ratio (UACR) of 300 mg/g or higher
4. History of acute kidney injury (AKI) during the 6 months prior to screening g.
5. Intolerance or allergy to Protality Base or Ensure Max Protein or to any of its ingredients
6. Women who are pregnant or lactating or expect to be pregnant or lactating during the study period.
7. Women of childbearing potential who are not using highly effective contraceptive methods.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in lean muscle mass from baseline | Endpoints will be analyzed at three months and six months.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hamdy, MD, PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided